CLINICAL TRIAL: NCT03960554
Title: The Effects of 12-months of Denosumab on Bone Density, Quality and Strength in Prevalent Kidney Transplant Recipients
Brief Title: The Effects of 12-months of Denosumab on Bone Density in Prevalent Kidney Transplant Recipients
Acronym: ProliaKTx
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study lost funding
Sponsor: Thomas Nickolas, MD MS (Other)
Responsible Party: Sponsor-Investigator, Thomas Nickolas, MD MS, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAS3103
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Osteoporosis; Renal Osteodystrophy; Kidney Transplant; Complications
Keywords: Denosumab; Bone density; Kidney transplant; Prolia
MeSH Terms: conditions — Osteoporosis; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigators and clinical research coordinators will be blinded to treatment assignment for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active drug (Active Comparator): Denosumab 60 mg subcutaneous injection every 6 months for 12 months (i.e., 2 injections)
  Interventions: Drug: Denosumab Inj 60 mg/ml
- Placebo (Placebo Comparator): Placebo subcutaneous injection every 6 months for 12 months (i.e., 2 injections)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Denosumab Inj 60 mg/ml — Treatment will be administered by study personnel as a subcutaneous injection every 6-months for one year.
  Other Names: Prolia
  Arms: Active drug
Other: Placebo — Placebo will be administered by study personnel as a subcutaneous injection every 6-months for one year.
  Arms: Placebo

SUMMARY:
This is a Phase 2 Multi-Center Clinical Trial (safety and effectiveness trial) in 60 patients (40 denosumab; 20 placebo) who have had a kidney transplant for 12-months or longer with more than 30% of kidney function. The investigators will test whether denosumab safely improves bone mineral density (BMD) by dual-energy X-ray absorptiometry (DXA) and improves bone strength by high resolution peripheral quantitative computed tomography (HR-pQCT) in the subset of patients recruited at Columbia University Irving Medical Center. These data will inform the development and execution of a larger trial to test if denosumab prevents fractures in kidney transplant recipients.

DETAILED DESCRIPTION:
Bone fractures are 3-times more common in kidney transplant recipients than in the general population and risk of dying after a hip fracture is 60% higher compared to kidney transplant recipients without a fracture. Unfortunately, there are no anti-fracture strategies that have been proven to be effective in double blinded randomized clinical trials for kidney transplant recipients. This is because some anti-fracture medications that are commonly used to treat osteoporosis and prevent fractures in the general population (i.e., bisphosphonates), may be harmful to the skeleton when kidney function is less than 30% of normal. In addition, intravenous bisphosphonates may be toxic to the kidneys, which further limits their utility in patients with a kidney transplant.

Denosumab, a monoclonal antibody against RANKL, inhibits osteoclast function and is not harmful to the kidney. Denosumab prevents fractures in men and women with age-related and glucocorticoid-induced osteoporosis. Recently, a non-blinded randomized trial of denosumab versus usual care during the first year of kidney transplantation in 90 patients reported the bone mineral density (BMD) measured by dual energy X-ray absorptiometry (DXA) increased at the spine and hip and that bone strength measured by high resolution peripheral quantitative computed tomography (HR-pQCT) increased in patients treated with denosumab. Adverse events in denosumab-treated patients included greater risk of urinary tract infections, diarrhea, and transient levels of low serum calcium that were asymptomatic. This study demonstrated that denosumab safely increased BMD at the spine and hip in new kidney transplant recipients. However, long-term kidney recipients, who comprise the vast majority of patients living with a transplanted kidney and who are also at increased risk of fracture, were not included.

ELIGIBILITY:
Inclusion criteria

1. Men and women
2. All race-ethnicities
3. Age ≥ 18 years
4. ≥ 12-months after kidney transplantation (living or deceased donor recipient)
5. Stable allograft function over the previous year defined as:

   1. No rejections
   2. No more than a 15% decline in Glomerular filtration rate (GFR) over the prior year
6. Allograft GFR ≥ 30 mL/minute/1.73 m2 (MDRD or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) per local lab reporting)
7. 25OHD ≥ 30 ng/mL (determined at screening visit)
8. Serum calcium ≥ 9.0 mg/dL (determined at screening visit)
9. T-Score at the spine including and between -1.0 and -3.5 (determined at screening visit)
10. Must have had a routine dental exam within 6-months of study recruitment
11. Must agree to continue with routine dental exams over the course of the study
12. Has not undergone an invasive dental procedure (i.e., tooth extraction, dental implants, oral surgery) within ≤ 3-months of recruitment
13. Must agree to referral to metabolic bone disease specialist at the end of the study
14. Women of child bearing potential must be willing to use one form of effective contraception over the course of the study

Exclusion Criteria

1. Allograft GFR < 30 mL/minute/1.73 m2 (MDRD or CKD-EPI per local lab reporting)
2. Within 24-months of starting renal replacement therapy
3. Prevalent or occult vertebral fractures
4. History of post-transplantation non-basal cell carcinoma cancers
5. Non-ambulatory
6. Malignancy requiring chemotherapy or metastatic to bone
7. Non-transplant related metabolic bone diseases that alter bone mineral density, including but not limited to Primary hyperparathyroidism, Paget's, Osteogenesis Imperfecta
8. Within one-year of parathyroidectomy
9. Untreated hyperthyroidism for 6-months or longer
10. Untreated hypothyroidism for 6-months of longer
11. Medical diseases (end stage liver, lung or heart, intestinal malabsorption)
12. Use within the prior year of bisphosphonates, teriparatide, selective estrogen receptor modulators, testosterone, estrogen, denosumab, abaloparatide, calcitonin, and romosozumab
13. Allergy to components within the denosumab preparation or to denosumab
14. Weight > 300 pounds
15. Parathyroid hormone (PTH) > 450 pg /mL
16. Will undergo an invasive dental procedure (i.e., tooth extraction, dental implants, oral surgery) within the next 12-months
17. Pregnant
18. Planned pregnancy during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nickolas, MD, MS, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Northwestern University, Feinburg School of Medicine, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Drug | Placebo
Started | 4 | 4
Completed | 0 | 0
Not Completed | 4 | 4
Not completed — Due to the pandemic, this study was terminated early | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD) Measured by Dual Energy X-ray Absorptiometry (DXA)
Description: BMD will be measured to determine if 1-year of treatment with denosumab changes BMD as measured by DXA.
Time Frame: 12 months
Population: Data was not collected due to termination of the study.
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Estimated Bone Strength Measured by High Resolution Peripheral Quantitative Computed Tomography (HR-pQCT) Imaging
Description: Estimated bone mechanical competence will be measured by HR-pQCT.
Time Frame: 12 months
Population: Data was not collected due to termination of the study.
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to one year
Arm/Group | Active Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Drug (N=4) | Placebo (N=4)
left elbow pain (Musculoskeletal and connective tissue disorders) | 0 | 1
cold sore (Skin and subcutaneous tissue disorders) | 0 | 1
Gastrointestinal Disorder (unspecified) (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, this study was terminated early and no Outcome Measure data was collected from participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03960554/Prot_SAP_000.pdf